CLINICAL TRIAL: NCT06040242
Title: Characterization of Arrhythmogenic Activity During and After Physical Exercise in Patients With Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Brief Title: Arrhythmogenic Activity During Exercise in ARVC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EAP_2020
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: exercise; cycling; physical activity
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Motor Activity | interventions — Exercise; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Group (Experimental): All patients will perform all exercises. Arrhythmogenic activity will compared with that assessed during treadmill walking.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will perform 3 min of the different activities, followed by a 10-min recovery window.
  Other Names: cycling, squats, biceps curls, walking

SUMMARY:
Current guidelines advocate that ARVC patients, typically young and active individuals with a significant history of competitive endurance sports, cease endurance training in favour of activities with low cardiac burden such as bowling and golf. Empirically, it is often suggested that heart rate during exercise should not exceed 100-120 bpm in these patients, but these guidelines are arbitrary and not scientifically based. In practice, it is estimated that up to 50% of patients do not comply with these recommendations .

Adequate quantification of the arrhythmogenic burden, defined as premature ventricular beats in proportion to all heart beats in each period of time, and cardiac load (defined as stroke volume for volume load and systolic blood pressure for pressure load) experienced by ARVC patients when performing different types of physical exercise would be a first step towards designing a safe and effective intervention so that these patients can profit from an active life style.

This study therefore aims to quantify and describe the arrhythmogenic burden and cardiac load experienced by patients with ARVC while performing different physical exercise over a range of intensities - all strictly within the range currently recommended by different cardiological societies.

DETAILED DESCRIPTION:
In this study, ARVC patients with different genotypes will perform a series of different physical activities, including treadmill walking, cycling at different intensities, biceps curls and loaded squats while undergoing extensive cardiovascular monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Definitive ARVC diagnosis according to the modified 2010 ARVC Task Force Criteria
* Pathogenic / likely pathogenic variant in one of the following desmosomal genes: plakophilin-2 (PKP-2), desmoglein-2 (DSG-2) or desmoplakin (DSP) or gene-elusive definite ARVC (i.e., genetic test performed but no pathogenic / likely pathogenic variant found)
* Agreement with responsible primary cardiologist that study participation is not considered beyond acceptable levels of physical activity for this particular patient
* No history of exercise-induced syncope in the 6 months prior to study participation
* No history of sudden cardiac arrest in the 6 months prior to study participation
* In patients who suffered from sudden cardiac arrest/arrhythmic syncope, only those having an implantable cardioverter-defibrillator (ICD) and being under beta-blockers/antiarrhythmic drugs are eligible for study inclusion
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age: > 18 years
* Body-Mass-Index (BMI): 18.5 - 29.9 kg･m-2
* Willing to adhere to the following study rules:

  * No intense exercise 48h prior to testing
  * No exercise 24h prior to testing
  * Sleep at least 7h the two nights before testing On test day
  * No caffeinated food or drink before testing on test day
  * No alcohol before testing on test day
  * Fully compliant with normal medication regimen including beta-blockers and antiarrhythmic medication

Exclusion Criteria:

* No genetic test history for ARVC variants
* Heart failure with severely reduced left ventricular ejection fraction (LVEF <35%)
* For women: Pregnancy, breastfeeding, or intention to become pregnant during the study.
* Known or suspected non-compliance, drug, or alcohol abuse
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
count of premature ventricular beats during and after the activities | measured during the 3 min of activity and the 10 min of recovery
  count of premature ventricular beats during and after the activities

SECONDARY OUTCOMES:
cardiac load during different activities, as rate-pressure product | measured during the 3 min of activity
  product of heart rate and systolic blood pressure
cardiac load during different activities, as cardiac output | measured during the 3 min of activity
  product of heart rate and stroke volume, in L/min
cardiac load during different activities, as peak blood pressure | measured during the 3 min of activity
  systolic blood pressure, in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Spengler, PhD, MD, Principal Investigator — ETH Zurich, Exercise Physiology Lab, Institute of Human Movement Sciences and Sport
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No